CLINICAL TRIAL: NCT07038889
Title: Investigating the Feasibility and Translational Therapeutic Benefits of Overground, Fully Immersive Virtual Reality (VR) Gait Rehabilitation Therapies for Individuals With Traumatic Brain Injury (TBI)
Brief Title: Overground Virtual Reality (VR) Gait Rehabilitation for Traumatic Brain Injury (TBI)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Indiana University Health (Other)
Responsible Party: Principal Investigator, Hee-Tae Jung, Assistant Professor, Health Informatics, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25423
Record Dates: First submitted 2025-06-10; First posted 2025-06-26 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Traumatic Brain Injury; Stroke; Gait Training
MeSH Terms: conditions — Brain Injuries, Traumatic; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- VR-Assisted Overground Gait Therapy (Experimental): Participants in the treatment group (VG-AOGT) will engage in gait training within a newly developed immersive virtual reality (VR) environment. This setup features self-propelled overground walking influenced by three different virtual environments designed to mimic real-world conditions. The immersive technology used is HTC VIVE Pro 2, enabling participants to practice walking in real-world environments and gait tasks.
  Interventions: Device: Walk-over-Ground
- Conventional Treadmill-Based VR Gait Therapy (Active Comparator): Participants in the control group (VR-CTGT) will engage in gait training using C-Mill VR+ technology, which involves treadmill-assisted walking on a treadmill while interacting with less immersive virtual scenarios presented on screens.
  Interventions: Device: C-Mill VR+ by Motek

INTERVENTIONS:
Device: C-Mill VR+ by Motek — Participants perform treadmill-assisted walking while interacting with non-immersive, game-like environments displayed on screens attached to the treadmill.
  Arms: Conventional Treadmill-Based VR Gait Therapy
Device: Walk-over-Ground — This intervention utilizes the HTC VIVE Pro 2 system for a realistic, fully immersive VR-assisted overground gait therapy. The immersive VR environment is designed to mimic real-world scenarios and challenges, enhancing the rehabilitation process by engaging patients in naturalistic gait activities.
  Arms: VR-Assisted Overground Gait Therapy

SUMMARY:
The purpose of this study is to evaluate a new virtual reality (VR)-based rehabilitation program designed to help individuals with traumatic brain injury (TBI) improve their walking abilities in real-world settings. By comparing immersive VR-assisted overground gait therapy to contemporary non-immersive, treadmill-based VR therapy (i.e., C-Mill), the investigators aim to determine its effectiveness in enhancing mobility and quality of life for TBI patients.

DETAILED DESCRIPTION:
After obtaining consent and screening, eligible participants are randomized to the treatment or control groups.

First, all participants are issued a wearable tracker to gauge baseline activity for at least 5 days.

During the intervention phase, participants undergo 12 treatment sessions, 2x a week for 6 weeks.

Assessments are conducted at pre-intervention, post-intervention, and 1-month followup.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: A confirmed diagnosis of traumatic brain injury (TBI) or stroke, confirmed by the referring neurologist.
* Cognitive Function: Mini-Mental State Examination (MMSE) score greater than 24, indicating sufficient cognitive function to participate in the study.
* Exercise Clearance: Approval from a neurologist for participation in exercise-based interventions.
* Rehabilitation Need: Demonstrates a need for functional rehabilitation.
* Recent Therapy: Participants should not have received physical therapy (PT) within the last month.
* Consent: Must be able to provide informed consent for themselves.

Exclusion Criteria:

* Participants with unstable medication regimens that could interfere with their participation in the study.
* Any comorbidity that could interfere with walking or gait training.
* Participation in VR-assisted gait training within the last 6 months.
* Intolerance to virtual reality environments or motion simulation.
* Severe cognitive, visual, or hearing impairments where the participant cannot follow the therapist's instructions.
* More than 135 kg total body weight.
* More than 2.00 meters in body height.
* Presence of open skin lesions or bandages in areas that would come into contact with the harness.
* Functional Ambulation Category (FAC): Participants with an FAC score of less than 2 indicate they require physical support from more than one person to walk.

Clarification:

- The diagnosis of TBI or stroke can be confirmed by their neurologist or a physical therapist referring to the patient. If a physical therapist makes the referral, the diagnosis must still be officially confirmed by a neurologist to ensure it meets the study's medical criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Step Count | Continuous tracking from Screening to Week 10
  FitBit tracks the number of steps (count) taken by participant.
Travel Distance | Continuous tracking from Screening to Week 10
  FitBit tracks the total distance (miles) travelled by participant.
Activity Zone Minutes | Continuous tracking from Screening to Week 10
  Fitbit calculates maximum heart rate (HR) from user age (Max HR = 220 - age) and defines Activity Zone thresholds based on percentages of max HR (Fat Burn 50-69%, Cardio/Peak >70%).
  Activity Zone Minutes (AZMs) are an intensity-weighted measure of activity. AZM (count) is based on sustained heart rate over time: 1 AZM per minute in the Fat Burn Zone (50-69% max HR) and 2 AZMs per minute in the Cardio/Peak Zones (>=70% max HR).

SECONDARY OUTCOMES:
10-Meter Walk Test | Baseline, Week 7, Week 10
  10MWT: Subjects will walk a distance of 10 meters at their normal pace while being timed, allowing assessment of gait speed and mobility. (5 minutes)
6-Minute Walk Test | Baseline, Week 7, Week 10
  6MWT: Subjects will walk for 6 minutes along a 30m track. Subjects may stop and rest as often as needed. Subject walking speed will be collected during the test to evaluate the rate of functional fatigue. (10 minutes)
Dynamic Gait Index | Baseline, Week 7, Week 10
  DGI: Subjects will complete 14 different tasks ranging from static standing to dynamic walking. All subjects will be guarded closely for safety to prevent falling. (15 minutes)
Timed Up and Go Test | Baseline, Week 7, Week 10
  TUG: Subjects will rise from a seated position, walk three meters, turn around, walk back to the chair, and sit down. This test is used to assess mobility, balance, walking ability, and fall risk. (5 minutes)
Step-Over Test | Baseline, Week 7, Week 10
  SOT: Patients will walk over a flat firm surface for 14 meters. The pathway will include a box that is one foot wide. Each participant will complete 10 passes, stepping over the obstacle (box) each time taking about 15 minutes.
Step Length | Baseline, Week 7, Week 10
  With the PKMAS Zeno Walkway (ProtoKinetics), participants walk over a 14-foot pressure mat to capture gait kinematics. Step length (centimeters) measures the distance between the heel contact point of one foot to the heel contact point of the other foot.
Stride Length | Baseline, Week 7, Week 10
  With the PKMAS Zeno Walkway (ProtoKinetics), participants walk over a 14-foot pressure mat to capture gait kinematics. Stride length (centimeters) measures the distance between successive heel contact points of the same foot.
Stance Percentage | Baseline, Week 7, Week 10
  With the PKMAS Zeno Walkway (ProtoKinetics), participants walk over a 14-foot pressure mat to capture gait kinematics. During the gait cycle, each foot alternates between being in contact with the ground (stance phase) and not in contact with the ground (swing phase). Stance percentage (percent) is the proportion of the gait cycle during which a foot remains in the stance phase.
Gait Speed | Baseline, Week 7, Week 10
  With the PKMAS Zeno Walkway (ProtoKinetics), participants walk over a 14-foot pressure mat to capture gait kinematics. Gait speed (meters per second) is calculated by dividing the distance walked (meters) by the time taken (seconds).

OTHER OUTCOMES:
Quality of Life after Brain Injury | Baseline, Week 7, Week 10
  QoLIBRI: Participants will complete a questionnaire assessing the health-related quality of life specifically tailored for individuals recovering from brain injury.
Disability Rating Scale | Screening, Baseline, Week 7, Week 10
  DRS: Participants will complete a questionnaire assessing the level of disability and functional impairment. NOTE: Only applicable to TBI participants.
Mini-Mental State Examination | Screening
  The Mini-Mental State Examination (MMSE) is an 11-question cognitive performance assessment that evaluates orientation, understanding, language, attention, and memory.

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Tae Jung, Ph.D., Principal Investigator — Indiana University, Luddy School of Informatics, Computing, and Engineering; Peter Altenburger, Ph.D., PT, Principal Investigator — Indiana University, School of Health & Human Sciences; Indiana University Health, Center for Advanced Neurorehabilitation
Locations (1):
- Indiana University Health, Neurorehabilitation & Robotics, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided